CLINICAL TRIAL: NCT06915883
Title: The Use of Experiential and Relaxation Virtual Reality to Minimize Anxiety in Children With Life-Limiting Conditions
Brief Title: Experiential and Relaxation Virtual Reality as a Tool for Easing Anxiety in Seriously Ill Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Collaborators: Motol University Hospital (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Anna Zubková, Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EK-670/24; 187724 (Other Grant/Funding Number: Charles University Grant Agency)
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Palliative Care; Life Limiting Conditions; Life Threatening Diseases
Keywords: experiential VR; relaxation VR; modern technologies in supportive care in medicine; pediatric palliative care; virtual reality; anxiety reduction; pediatric

STUDY DESIGN:
Intervention Model Description: Two virtual reality interventions (experiential and relaxation) are provided to subjects at different time periods, the sequence of treatments is randomized for each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM 1: relaxation VR followed by experiential VR (Experimental)
  Interventions: Device: Relaxation virtual reality (VR); Device: Experiential virtual reality (VR)
- ARM 2: experiential VR followed by relaxation VR (Experimental)
  Interventions: Device: Relaxation virtual reality (VR); Device: Experiential virtual reality (VR)

INTERVENTIONS:
Device: Relaxation virtual reality (VR) — A newly developed self-guided app BreezeTrerraVR that helps patients practice relaxation breathing in an immersive virtual environment, using voice prompts, visual cues, and respiratory biofeedback for guidance. The app was developed in the VR center at the National Institute of Mental Health, Czech Republic (supported by THE JOHANNES AMOS COMENIUS PROGRAMME (OP JAC) EXCELLENCE IN RESEARCH, Title: Research of Excellence on Digital Technologies and Wellbeing, Project Registration Number: CZ. 02.01.01/00/22_008/0004583).
Device: Experiential virtual reality (VR) — The experiential VR intervention will use the VR program "Ocean Rift" (an experience of the underwater world and its animals). It is a calm experiential and distraction game program that does not require much mobility and interaction and is therefore suitable for pediatric patients and hospital environments. This VR application is also used in available published research.

SUMMARY:
The goal of this clinical trial is to assess the use of experiential and relaxation virtual reality (VR) interventions in easing anxiety and other distress symptoms in children with life-limiting and/or life-threatening conditions (LLC/LTC). The main questions it aims to answer are:

1. Does experiential and relaxation VR help to decrease anxiety in severely ill children?
2. What effect does it have on pain and fear?
3. Is there a difference between experiential and relaxation VR in the observed outcome measures?
4. How is the newly developed relaxation VR app BreezeTerraVR perceived by children with LLC/LTC?
5. How do caregivers of the patients perceive VR as an intervention tool for psychological distress? Researchers will compare baseline levels of outcome measures (e.g. anxiety) to post-intervention levels to determine if there is an effect.

Participants will:

* Experience both types of VR interventions-experiential and relaxation VR-for 7 to 15 minutes in two sessions (the number of days between sessions will depend on each child's medical plan), the order of interventions is randomized.
* Fill out a set of short questionnaires before and after each intervention (approximately 5 minutes per phase).

ELIGIBILITY:
Inclusion Criteria:

* age 7-17.9 years
* sufficient level of contact with the environment and ability to cooperate
* children and parents fluent in Czech
* diagnosis of a life-threatening or life-limiting disease according to the internationally accepted list of palliatively relevant diagnoses
* pediatric patients treated at the University Hospital Motol

Exclusion Criteria:

* age below 7 or above 17.9 years
* unstable health status
* inability to speak Czech
* absence of parental consent for participation in the study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety Levels from Baseline following Experiential and Relaxation Virtual Reality Intervention. | Baseline and 15 minutes (post intervention).
  Anxiety levels are always measured pre- and post- both VR interventions (relaxation and experiential) using a standardized Czech scale called the "Scale Measuring Anxiety in Children". The scale consists of 17 items, each rated on a 1-4 scale; however, only 15 items are included in the final score. The total score thus ranges from a minimum of 15 to a maximum of 60, with higher scores indicating higher levels of anxiety. The difference between baseline and post-intervention scores is then calculated
Feasibility and Acceptability of the Relaxation App in Pediatric Population. | 3-5 minutes post VR intervention
  The relaxation VR app is newly developed and has so far been tested only in adult populations. To measure its feasibility and acceptability, the Simulation Sickness Questionnaire (SSQ), two items from the System Usability Scale (SUS), and several non-standardized questions assessing levels of immersion, enjoyment, engagement, relaxation, and distraction will be used. These scales and items are administered post-intervention.
  The SSQ consists of 16 items rated on a 0-3 scale, with a total score range from 0 to 48; higher scores indicate a higher level of simulation sickness. The SUS items use a 1-5 scale (1 = totally agree, 5 = totally disagree), where lower scores reflect better usability. The non-standardized questions also use a 1-5 scale (1 = totally agree, 5 = totally disagree), with lower scores indicating higher levels of immersion, enjoyment, engagement, relaxation, and distraction.

SECONDARY OUTCOMES:
Change in Pain Levels from Baseline following Experiential and Relaxation Virtual Reality Intervention. | Baseline and 15 minutes (post intervention).
  To measure pain levels, the Wong-Baker Faces Pain Rating Scale is used. It is a 1-item scale designed to assess pain among pediatric patients, with scores ranging from 0 to 10. The scale is administered pre- and post-intervention. A higher score indicates a higher level of pain, with 0 representing no pain and 10 representing the most severe pain.
Change in Fear Levels from Baseline following Experiential and Relaxation Virtual Reality Intervention. | Baseline and 15 minutes (post intervention).
  To measure fear levels, the Child Fear Scale is employed. It is a 1-item visual scale designed to assess fear associated with medical procedures and hospitalization. The scale ranges from 0 to 4, with higher scores indicating higher levels of fear. It is administered at baseline (pre) and post-intervention, with 0 representing no fear and 4 indicating the highest level of fear.

OTHER OUTCOMES:
Parents' Opinion on the VR Relaxation and Experiential Interventions for Children/Child Patients. | From enrollement of the child to the end of second session (approximately 4 weeks from enrollement).
  Verbal opend-ended question on how the caregivers of the child patient perceive the VR intervention. This outcome is analysed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Fajnerova, MSc, PhD, Study Chair — National Institute of Mental Health (NIMH)
Locations (1):
- University Hospital Motol, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in respect to the outcome measures (baseline and post-treatment), meaning pre-processed data of individuals related to the study's outcome measures. All data will be anonymized, with each participant's data stored under a unique individual code.
Time Frame: IPD will be shared upon request once the entire project is completed and the study is published in a peer-reviewed impact journal in open-access mode.
Access Criteria: The IPD can be accessed by anyone upon request to the authors of the study. The authors can be contacted via email, which will be provided in the study publication and on the registration website.

REFERENCES:
- [Background] Toman J. Škály na měření úzkosti a úzkostlivosti u dětí. Praha: Národní ústav pro vzdělávání; 2018.
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Kennedy R, Lane N, Berbaum K, Lilienthal M. Simulator Sickness Questionnaire: An enhanced method for quantifying simulator sickness. Int J Aviat Psychol. 1993;3(3):203-20.
- [Background] Gerceker GO, Bektas M, Aydinok Y, Oren H, Ellidokuz H, Olgun N. The effect of virtual reality on pain, fear, and anxiety during access of a port with huber needle in pediatric hematology-oncology patients: Randomized controlled trial. Eur J Oncol Nurs. 2021 Feb;50:101886. doi: 10.1016/j.ejon.2020.101886. Epub 2020 Dec 1. PMID 33321461
- [Background] Fraser LK, Gibson-Smith D, Jarvis S, Norman P, Parslow R. 'Make Every Child Count' Estimating current and future prevalence of children and young people with life-limiting conditions in the United Kingdom FINAL REPORT FEBRUARY 2020. 2020;(February):1-61
- [Background] Foundation WBF. Wong-Baker FACES® Pain Rating Scale. 2016.
- [Background] Caruso TJ, George A, Menendez M, De Souza E, Khoury M, Kist MN, Rodriguez ST. Virtual reality during pediatric vascular access: A pragmatic, prospective randomized, controlled trial. Paediatr Anaesth. 2020 Feb;30(2):116-123. doi: 10.1111/pan.13778. Epub 2019 Dec 19. PMID 31785015